CLINICAL TRIAL: NCT06063031
Title: Investigation of a Specialized Nutritional Intervention and Rehabilitation Treatment in Patients With Post-COVID Condition to Improve Their Quality of Life: ARACOV-02
Brief Title: Nutritional Intervention and Rehabilitation Treatment in Patients With Post-COVID Condition
Acronym: ARACOV-02
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Instituto de Investigación Sanitaria Aragón (Other)
Collaborators: Solutex GC S.L. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: C.I. PI22/335
Record Dates: First submitted 2023-09-27; First posted 2023-10-02 (Actual); Last update posted 2024-11-15 (Actual); Status verified 2024-01

CONDITIONS: Post-COVID Condition
Keywords: Fatigue; Telerehabilitation; Functional Status; Physical Therapy; Nutrition Supplement; Multimodal Program; Quality of Life; Psychosocial factors; Anxiety; Depression
MeSH Terms: conditions — Post-Acute COVID-19 Syndrome; Fatigue; Anxiety Disorders; Depression | interventions — Exercise

STUDY DESIGN:
Intervention Model Description: Prospective, multicentric, double-blind randomized clinical trial
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Active nutritional supplement plus telerehabilitation (Experimental): Active nutritional supplement plus telerehabilitation
  Interventions: Dietary Supplement: Active
- Placebo nutritional supplement plus telerehabilitation (Placebo Comparator): Placebo nutritional supplement plus telerehabilitation
  Interventions: Other: Placebo

INTERVENTIONS:
Dietary Supplement: Active — Active nutritional supplement plus telerehabilitation
  Arms: Active nutritional supplement plus telerehabilitation
Other: Placebo — Placebo nutritional supplement plus telerehabilitation
  Arms: Placebo nutritional supplement plus telerehabilitation

SUMMARY:
SARS-CoV-2 is the coronavirus responsible for developing the disease known as COVID-19. Once the acute phase of the disease has passed, about 40% of the people who discharged continue to have symptoms, and of these, between 50 and 70% present them up to three months later. These persistent symptoms include physical aspects such as fatigue and dyspnea, but also cardiac such as palpitations, cognitive such as mental confusion, and psycho-emotional such as depression, anxiety, and stress. SARS-CoV-2 infection is associated with a hyperinflammatory state, including excessive inflammatory cell infiltration, inflammasomes activation. In this context, omega-3 metabolites (Special Pro-resolving Mediators-SPMs) restore the balance in nutritional and molecular levels of eicosanoids. A more direct and targeted way to increase SPMs levels is Omega3 Essential Nutrition with natural SPMs taken by mouth. Today, there are dietary supplements containing SPMs (LIPINOVA®), made from fish oil through a fractionation process. LIPINOVA® is a nutritional supplement patented by Solutex GC S.L., obtained through several fractionation stages (extraction, purification, separation, concentration) from rich-in-omega-3 fish oil (without additives). Each capsule contains 498 mg of fish oil and 2 mg of tocopherols. This represents a variable quantity from 50 to 150 mg of EPA (20%), a variable quantity from 100 to 225 mg of DHA (30%), as well as the following quantities of EPA and DHA active metabolites, obtained from a pool of natural lipid mediators contained in omega-3 oil: 40-200 mcg of 17-HDHA, 25-200 mcg of 18-HEPE and 20-100 mcg of 14-HDHA.

In addition to this, the appearance of this new health condition, post-COVID condition, has once again led physiotherapists to update themselves in search of the best evidence to guide the examination and necessary rehabilitation interventions in this type of patient. Studies have shown how physiotherapy sessions that include a multimodal program could be the most indicated for this type of patients. Patients with this condition present an increase in fatigue, dyspnea and a decrease in their functional capacity and, therefore, a decrease in their quality of life, due to various pathogenic mechanisms that include chronic hyperinflammation.

These patients could obtain greater health improvements in terms of their quality of life if a therapeutical exercise and education program based on tele-rehabilitation is implemented together with a natural nutritional supplement that generates a systemic anti-inflammatory effect through SPMs (omega- 3).

DETAILED DESCRIPTION:
Patients who have contracted COVID-19 usually show various symptoms during the infection: Fever, cough, generalized pain, gastrointestinal disturbances, dyspnea, and fatigue. The latter two symptoms occur in about half of patients worldwide, although they are even more common in Europe. In addition to these respiratory symptoms, the disease can also have effects at the muscular, neurological, and cardiovascular levels.

After the acute phase of the disease, approximately 40% of discharged patients still have symptoms, and of these, 50% to 70% have symptoms up to three months later. These persistent symptoms include physical aspects such as fatigue and shortness of breath, but also cardiac symptoms such as palpitations, cognitive symptoms such as mental confusion, and psychoemotional symptoms such as depression, anxiety, and stress.

However, it is also observed how this clinic can be maintained beyond three months. It is known that there is a group of patients, about 5-10%, who have persistent symptoms over a period of up to 2 years, and new symptoms may even appear, leading to persistent COVID. Although the terminology for designating patients with this persistent clinical condition is changing, on October 6, 2021, the WHO published a consensus document defining the post-COVID condition (CPCOVID).

The possible mechanisms contributing to the overall pathophysiology of CPCOVID are still unclear, and numerous factors have been proposed to date. A key element may be the presence of a state of chronic hyperinflammation. In the lung context, the virus activates innate immunity, leading to a cascade of inflammatory cytokines, including interleukin-6 (IL -6), IL -1, tumor necrosis factor-alpha, and reactive oxygen species. Some studies have attempted to demonstrate the presence of T cells and NK lymphocytes in these patients, making it appear that COVID is characterized by alterations in TCD4+ cells and TCD8+ cells.

Other proposed mechanisms include autoimmune mechanisms through the presence of autoantibodies that act against modulatory proteins that alter immune function. Also, the hypercoagulable state (thromboinflammatory state) associated with SARS-CoV-2 infection is responsible for the disproportionately high rates (20-30%) of thrombotic complications observed in patients with COVID-19 and autonomic nervous system involvement leading to autonomic dysfunction.

Therefore, controlling systemic inflammation and eliminating it in general is as important as eradicating the virus itself. In particular, omega-3 fatty acids (EPA and DHA) are substrates that modulate the immune system response by promoting the resolution of inflammation by producing pro-resolving mediators that actively modulate and resolve the immune system response. Thus, omega-6 (ARA) and omega-3 fatty acids (EPA and DHA) are structural lipids, but the biological effects are carried out by their naturally produced metabolites (SPMs). In cases where the acute response of the immune system is chronic, deficiency of SPMs in the affected tissues has been observed (e.g., in metabolic diseases {obesity, metabolic syndrome, diabetes type II, fatty liver}, dry eye, atherosclerosis, autoimmune diseases, etc.). These effects on the metabolic pathways of SPM production may reduce resolution and thus contribute to the chronicity of the inflammatory response.

Recently, severe COVID-19 was shown to be associated with an altered profile of SPMs compared with healthy individuals. SPMs may have a new role in the essential nutritional management of deficiencies of these metabolites in COVID-19 disease.

Several recent articles have suggested that the change in prostaglandin profile and the increase in arachidonic acid derivatives may be indicative of the severity of the disease and the chances of recovery in the patient with COVID-19.

In addition, the emergence of this new health condition, CPCOVID, has prompted physiotherapists to renew their search for the best evidence to guide the investigative and rehabilitative interventions required for this type of patient. Evidence is currently sparse, but it is known that cognitive function and emotional health are aspects that need to be considered in the patient's treatment plan, as well as the dynamics of general condition (weakness, fatigue, concentration, dizziness, headaches, sleep disturbances), anxiety, debilitating symptoms of decreased aerobic tolerance, and subjective feelings of severity of asthenia (fatigue, physical and mental tiredness, decreased motivation and activity). Studies have shown that physical therapy sessions that include: aerobic exercise, resistance aerobic exercise, strengthening exercises, diaphragmatic breathing techniques, and mindfulness training are most appropriate for this type of patient. Moreover, the use of new information and communication technologies (digital health) for rehabilitation treatment has also proven effective for other diseases such as cardiac, neurological, respiratory or musculoskeletal disorders.

Objective: To evaluate the improvement in quality of life in CPCOVID patients after a 12-week specialized nutritional intervention with (natural and standardized SPMs nutritional supplement) together with a therapeutic exercise and education program via telerehabilitation compared to a group that underwent the tele-rehabilitation program and no supplements (placebo), as measured by the Quality of Life Scale ( EQ-5D).

ELIGIBILITY:
Inclusion Criteria:

* To have signed the informed consent form.
* Age between 18 and 70 years with access to and knowledge of basic use of technological applications.
* Patients with clinical criteria of having suffered from COVID-19 with diagnosis confirmed by diagnostic techniques and systems in health centers (PCR, rapid antigen test, and/or serology (positive anti-N antibodies).
* Patients who remain symptomatic for more than 12 weeks after the onset of symptoms.
* Patients who manifest symptoms compatible with CPCOVID since the end of the acute phase*.
* Patients with fatigue greater than or equal to an average of 4 points on the FSS.
* Independent ambulation, even with the use of technical aids.

Exclusion Criteria:

* Patients with severe neurological diseases at the central and/or peripheral level that prevent them from following the program.
* Patients with respiratory insufficiency: SaO2 < 90% or respiratory rate ≧30.
* Patients with rheumatic diseases or acute musculoskeletal injuries that do not allow exercise.
* Patients who do not have access to the Internet or are unable to use the Internet on a daily basis.
* Patients with clinical symptoms consistent with chronic fatigue syndrome.
* Presence of symptoms consistent with CPCOVID prior to SARS Cov-2 infection.
* Pregnant or lactating women or women of childbearing age who are trying to become pregnant.
* Patients unable to follow oral and written instructions in Spanish.
* Patients with an allergy to fish, shellfish, or any of the ingredients of the preparation.
* Patients enrolled in another clinical trial for the treatment of symptomatology derived from COVID -19.
* Patients who have completed another clinical trial in the 4 weeks prior to enrollment.
* Patients who have received immunosuppressive medications and/or corticosteroids in the last 2 weeks prior to enrollment. Patients who have received nonsteroidal anti-inflammatory drugs (NSAIDs) continuously or on a fixed regimen in the 2 weeks prior to treatment initiation. Patients who have been taking NSAIDs may have a 7-day withdrawal period.
* Women of childbearing age who are not willing to take NSAIDs should not be treated.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 146 (Actual)
Dates: Start 2022-09-26 (Actual); Primary Completion 2025-01-15 (Estimated); Study Completion 2025-04-30 (Estimated)

PRIMARY OUTCOMES:
Changes in the Quality of life (EQ-5D) | Pre-intervention (day 1); after intervention (12 weeks)
  The EQ-5D is a generic instrument for measuring health-related quality of life that can be used in relatively healthy individuals (general population) as well as in patient groups with various medical conditions. Individuals rate their own health status, first in severity by dimension (descriptive system) and then on a more general visual analog scale (VAS). A third element of the EQ-5D is the index of social values, which is determined for each health status identified by the instrument. The descriptive system contains five health dimensions (mobility, self-care, activities of daily living, pain/discomfort, and anxiety/depression), each with five severity levels (no problems, mild problems, some problems or moderate problems, and severe problems, cannot occur). In each dimension of the EQ -5D, the severity levels are each coded from 1 to 5.

SECONDARY OUTCOMES:
Changes in the Biomarkers | Pre-intervention (day 1); after intervention (12 weeks)
  Cytokines: IL-1, IL-2, IL-6, IL8, IL10, IL17 TNF-α, IFNγ. Fatty acids: EPA, DHA, ARA, DPA. Monohydroxylated SPMs: 17-HDHA, 18-HEPE, 14-HDHA. Resolvins: RvE1, RvD1, RvD2, RvD3, RvD4, RvD5. Maresins: MaR1, MaR2. Proteins: PD1, PDX. Lipoxins: LXA4, LXB4. Prostaglandins: PGE2, PGD2, PGF2α. Thromboxanes: TXB2. Leukotrienes: LTB4
Changes in the Fatigue Severity Scale (FSS) | Pre-intervention (day 1); after intervention (12 weeks)
  The FSS is a self-assessment scale consisting of 9 items that relate fatigue severity to daily activities. Each item is scored on a scale of 1 to 7, from 1=disagree at all to 7=agree completely. An average of less than 3 points is considered no fatigue, less than 4 is considered mild fatigue, and 4 or more is considered severe fatigue. An average of 4 points is usually used as the cutoff point. This range can be divided into three fatigue blocks: 4 < 5= mild fatigue; 5 < 6= moderate fatigue; 6-7= very severe fatigue.
Changes in the Modified Medical Research Council Scale (mMRC) | Pre-intervention (day 1); after intervention (12 weeks)
  This scale can be used to determine the extent of dyspnea reported by the patient by using a scale from 0=no dyspnea to 4=does not leave the house because of dyspnea.
Changes in the Measurements of peak inspiratory pressure and peak expiratory pressure | Pre-intervention (day 1); after intervention (12 weeks)
  Peak inspiratory pressure is the pressure generated against a closed system at maximum inspiratory effort. It is usually measured by residual volume (RV) because inspiratory muscle force is inversely related to lung volume (in a curvilinear fashion). Peak expiratory pressure is measured during a similar maneuver using total lung capacity (TLC), since expiratory muscle force is directly related to lung volume (also in a curvilinear fashion). However, the information available on these maneuvers is nonspecific and does not allow discrimination between insufficient effort, muscle weakness, and a neurological disorder.
Changes in the Functional capacity as measured by the 6-minute walk | Pre-intervention (day 1); after intervention (12 weeks)
  Study participants must walk the maximum possible distance for 6 minutes. During walking, patients may rest if they wish. They are monitored with a pulse oximeter and follow the instructions of the physical therapist. The distance is measured in meters. The total distance walked by the participants is related to the distance estimated for their age, sex, height and person according to the Troosters equation.
Changes in the Functional capacity as measured by the 30-second sit-stand test | Pre-intervention (day 1); after intervention (12 weeks)
  This test should be performed on a chair high enough for the feet to rest on the floor. The patient's arms should be crossed in front of the chest. He should rise in this position and return to the starting position as many times as possible within 30 seconds. The total number of repetitions is compared to the estimated number of repetitions for each gender and age to determine who has normal or below average values.
Changes in the Functional capacity as measured by the 30-second elbow flexion test | Pre-intervention (day 1); after intervention (12 weeks)
  From a sitting position, the dominant arm should be used to perform as many bending and extending movements of the elbow as possible in 30 seconds with a weight of 2 kg for women and 4 kg for men.
Changes in the Psychosocial factors (anxiety severity) | Pre-intervention (day 1); after intervention (12 weeks)
  Overall Anxiety Severity and Impairment Scale (OASIS). Consists of five items that measure the frequency and severity of anxiety, as well as level of avoidance, work/school/home interference, and social interference associated with anxiety. The instructions orient the respondent to consider a wide range of anxiety symptoms (e.g., panic attacks, worries, flashbacks) when answering the questions, and the time frame is "over the past week." Respondents select among five different response options for each item, which are coded 0-4 and summed to obtain a total score. A psychometric analysis of the OASIS suggested that the scale was unidimensional and had good internal consistency, test-retest reliability, and convergent/discriminant validity (Norman et al., 2006).
Changes in the Psychosocial factors (depression severity) | Pre-intervention (day 1); after intervention (12 weeks)
  Overall Depression Severity and Impairment Scale (ODSIS). Consists of five items. This self-report assesses the severity and impairment of depressive symptoms and their interference with work, school, and social life. Of the five response options offered for each item, the person must select the one that best describes his or her symptoms. the person must select the one that best describes his or her experiences in the past week. The responses are coded on a scale of 0 to 4 and summed to give a total score of 0 to 20.
Measurement of the Adherence to the tele-rehabilitation program | Every 2 weeks, during 12 weeks of intervention.
  Adherence to the tele-rehabilitation program will be recorded.
Measurement of the Adherence to the Nutritional supplementation | Adherence: weeks: 2, 6 and 10 - % compliance: after intervention (12 weeks)
  Adherence to the nutritional supplement will be recorded.
  Moreover, the return of the nutritional supplement will also be taken into account. The patient will be asked if he/she has returned the remaining amount of nutritional supplement after completing the 12-week treatment. The following will be taken into account: the number of capsules taken; the number of capsules returned; and the number of capsules to be taken (336 for patients who have completed the 12 weeks. It should be indicated here if there have been any discontinued patients for whom the number of capsules that should have been taken would be calculated). From these data, the % compliance with the treatment with the medicine/nutritional supplement (by dividing the number of capsules taken by the number of capsules applicable to take and multiplying by 100) should be extracted.

OTHER OUTCOMES:
Clinical parameters and Socio-demographic data | Pre-intervention (day 1)
  Weight; height; BMI (clinical parameters) / Age; Gender; Race; Educational level; Cohabitation status; Profession (socio-demographic data)

CONTACTS AND LOCATIONS:
Overall Officials: Jorge Alamillo Salas, Dr, Principal Investigator — SALUD; Sandra Calvo Carrión., Dr, Principal Investigator — Universidad de Zaragoza; Beatriz Carpallo Porcar, MSc, Principal Investigator — Universidad San Jorge; Carolina Jiménez Sánchez, Dr, Principal Investigator — Universidad San Jorge; Ana Isabel Aller Blanco, Dr, Principal Investigator — SALUD; Elena Kolesnyk Sumskaya, Dr, Principal Investigator — SALUD; Esther del Corral Beamonte, Dr, Study Chair — SALUD; Pablo Herrero Gallego, Dr, Principal Investigator — Universidad de Zaragoza
Locations (1):
- IIS Aragón, Zaragoza, Spain

REFERENCES:
- [Derived] Carpallo-Porcar B, Jimenez-Sanchez C, Calvo S, Irun P, Kolesnyk-Sumskaya E, Aller-Blanco AI, Beamonte EDC. ARACOV-02. Specialized nutritional intervention and telerehabilitation in patients with long COVID: Protocol of a randomized controlled trial. PLoS One. 2025 Apr 29;20(4):e0321811. doi: 10.1371/journal.pone.0321811. eCollection 2025. PMID 40299883